CLINICAL TRIAL: NCT02187991
Title: A Phase II, Multicenter, Randomized, Parallel Group Study to Compare Alisertib in Combination With Paclitaxel vs. Paclitaxel Alone in Patients With Metastatic or Locally Recurrent Breast Cancer
Brief Title: Study to Compare Alisertib With Paclitaxel vs. Paclitaxel Alone in Metastatic or Locally Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-033
Record Dates: First submitted 2014-07-06; First posted 2014-07-11 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Tumors; Malignant Neoplasm of Breast
Keywords: metastatic breast cancer; Human Epidermal Growth Factor Receptor 2-negative (HER2-) breast cancer; Estrogen Receptor-positive (ER+) breast cancer; Triple Negative breast cancer; alisertib; paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Paclitaxel; Albumin-Bound Paclitaxel; MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ER+/HER2- Paclitaxel Alone (Active Comparator): Paclitaxel 90 mg/m2 IV on days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Paclitaxel
- ER+/HER2- Paclitaxel plus Alisertib (Experimental): Paclitaxel 60 mg/m2 intravenously (IV) on days 1, 8 and 15 of a 28-day cycle; Alisertib 40 mg twice a day (BID) on days 1-3, 8-10, and 15-17 of a 28-day cycle
  Interventions: Drug: Paclitaxel; Drug: Alisertib
- Triple Negative Paclitaxel Alone (Active Comparator): Paclitaxel 90 mg/m2 IV on days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Paclitaxel
- Triple Negative Paclitaxel plus Alisertib (Experimental): Paclitaxel 60 mg/m2 intravenously (IV) on days 1, 8 and 15 of a 28-day cycle; Alisertib 40 mg BID on days 1-3, 8-10, and 15-17 of a 28-day cycle
  Interventions: Drug: Paclitaxel; Drug: Alisertib

INTERVENTIONS:
Drug: Paclitaxel — either 60 mg/m2 intravenously (IV) on days 1, 8 and 15 of a 28-day cycle (on Paclitaxel plus Alisertib arm) or 90 mg/m2 IV on days 1, 8 and 15 of a 28-day cycle (on Paclitaxel Alone arm)
  Other Names: Taxol; Abraxane
Drug: Alisertib — 40 mg BID (twice a day) on days 1-3, 8-10, and 15-17 of a 28-day cycle
  Other Names: MLN8237
  Arms: ER+/HER2- Paclitaxel plus Alisertib; Triple Negative Paclitaxel plus Alisertib

SUMMARY:
The goal of this clinical research study is to learn if the study drug, alisertib (MLN8237), in combination with chemotherapy (paclitaxel), can shrink or slow tumor growth in women with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative or HR-negative, HER2-negative (triple negative) locally recurrent or metastatic breast cancer (MBC). The safety of alisertib in combination with paclitaxel will also be studied. The physical state of the patient, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if alisertib plus paclitaxel is safe and effective in patients with this type of breast cancer.

Alisertib belongs to a group of drugs called Aurora kinase inhibitors. Alisertib blocks the activity of Aurora A kinase, a protein that is involved in tumor cell multiplication and survival. Aurora A kinase is expressed at higher than normal levels in many types of cancer, including breast cancer, and preclinical studies suggest that blocking the activity of this protein can lead to the death of cancer cells.

Paclitaxel is a chemotherapy drug commonly used to treat many different kinds of cancer, including metastatic breast cancer. The reason to combine alisertib and paclitaxel is that in cancer therapy, combinations of drugs are often more effective as a treatment than either of the same drugs used alone.

DETAILED DESCRIPTION:
The rationale behind assessing the effectiveness of the addition of alisertib to weekly paclitaxel therapy in patients with Triple Negative Breast Cancer and highly proliferative estrogen receptor-positive (ER+) and HER2- breast cancer is based on the unmet clinical need for effective strategies to prevent or delay resistance to taxane therapy in the metastatic setting. Synergistic or additive effects have been observed in breast cancer xenograft models which involved alisertib added to either paclitaxel or docetaxel. Alisertib inhibited the Pgp-mediated efflux of paclitaxel in a cell culture model. In addition, Aurora Kinase A is frequently overexpressed in Triple Negative Breast Cancer (TNBC), and expression levels have been shown to be prognostic in both of these breast cancer subtypes. The combination of alisertib with paclitaxel has also been investigated in a Phase 1 study in patients with locally advanced or metastatic ovarian and breast cancers, with preliminary evidence of activity in both tumor types including 6 partial response (PR)s and 3 stable disease (SD) in 11 patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care, and signed Health Insurance Portability and Accountability Act (HIPAA) form.
* Female subject (≥18 years old), who is either:

  * post-menopausal for at least one year before the screening visit, or
  * surgically sterilized, or
  * willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide) for the duration of the study.
* Metastatic or locally recurrent breast cancer with histologic confirmation (on either primary or metastatic tumor) of one of the following:

  * ER+, HER2- invasive breast cancer (any progesterone receptor [PgR] status)
  * Poorly differentiated and/or Grade 3 invasive TNBC, defined as:
  * HER2 negative status (based on most recently analyzed biopsy) is defined as immunohistochemistry (IHC) status of 0, 1+ or 2+ (if IHC 2+, a negative FISH test is required, i.e., HER2 fluorescence in situ hybridization (FISH) ratio < 2.0 with an average HER2 copy number <4.0 signals/cell); ER-negative and PR-negative status is defined as ER and PgR <1% nuclei positive by IHC
* Measurable disease by modified Response Evaluation Criteria in Solid Tumors (RECIST) (v1.1) or non-measurable lytic, bone-only disease (mixed blastic/lytic bone disease is allowed); if patient has bone-predominant disease with no measurable disease, there must be a lytic component to the bone metastases that is visible on plain X-ray or CT scan that can be serially followed
* Absolute neutrophil count (ANC) > 1500/mm³, platelets > 100,000/mm³, Hgb > 9 g/dL. Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days, however, erythrocyte growth factor is allowed as per published American Society of Clinical Oncology (ASCO) guidelines (available at: http://www.asco.org/quality-guidelines/asco-ash-clinical-practice-guideline-update-use-epoetin-and-darbepoetin-adult).
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN), serum glutamic-oxaloacetic transaminase (SGOT) (AST) and serum glutamic-pyruvic transaminase (SGPT) (ALT) < 2.5 x ULN. AST and/or ALT may be up to 5 x ULN if patient has known liver metastases
* Adequate renal function as defined by: Calculated creatinine clearance must be ≥ 30 mL/minute (see Cockcroft-Gault formula in Appendix 5)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (refer to Appendix 4)

Exclusion Criteria:

* Previous radiation therapy covering the whole pelvis
* Suspected brain metastases, untreated brain metastases or current clinical or radiologic progression of known brain metastases or requirement for steroid therapy for brain metastases

  * Patients with treated brain metastases are eligible if they have been stable and off steroids for ≥ 3 weeks
* Prior allogeneic bone marrow or organ transplantation
* Known GI disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib. Examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen.
* Requirement for administration of proton pump inhibitor, or for constant administration of H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids or H2 antagonists are allowed as described in Section 3.4.
* Systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 3), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Female subject who is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening, within 72 hours prior to first dose of study drug(s). Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received an investigational agent within 30 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Other severe acute or chronic medical and/or psychiatric condition(s), including but not limited to uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormalities that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient not eligible for enrollment for this study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, or an in situ malignancy, or a stage I cancer with a 5-year Disease Free Survival (DFS) of ≥ 90% (survival rates by stage are available for most cancers on the American Cancer Society website).
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib and during the study.
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion. For guidance in defining active infection for hepatitis B, please refer to the World Health Organization (WHO) guidelines, Global Alert and Response (GAR), Hepatitis B. http://who.int/csr/disease/hepatitis/whocdscsrlyo20022/en/index4.html)
* Prior administration of an Aurora A kinase-targeted agent, including alisertib
* Need for ongoing therapeutic steroid therapy. Intermittent steroid use for the control of nausea and vomiting is allowed. Premedication with dexamethasone prior to paclitaxel administration is allowed. Topical steroid use is permitted. Inhaled steroids are permitted. Replacement doses of hydrocortisone up to 15 mg/day are allowed.
* Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to alisertib.
* Administration of myeloid growth factors or platelet transfusion within 14 days prior to the first dose of study treatment.
* More than 1 previous chemotherapy regimen for metastatic disease

  * No limit on previous endocrine therapy
  * Previous mammalian target of rapamycin (mTOR) therapy, e.g., everolimus, is allowed
  * Prior adjuvant taxane therapy is allowed, provided the disease-free interval from the end of (neo)adjuvant chemotherapy to the development of metastatic disease was ≥ 1 year
  * No prior taxane for metastatic disease
* Peripheral neuropathy > grade 1
* Known severe hypersensitivity to paclitaxel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A. O'Shaughnessy, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 22 Sites, Including Dallas and Austin, Texas, United States

REFERENCES:
- [Derived] O'Shaughnessy J, McIntyre K, Wilks S, Ma L, Block M, Andorsky D, Danso M, Locke T, Scales A, Wang Y. Efficacy and Safety of Weekly Paclitaxel With or Without Oral Alisertib in Patients With Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e214103. doi: 10.1001/jamanetworkopen.2021.4103. PMID 33877311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2015 and February 2018, a total of 169* women were enrolled in the trial and were randomly assigned to paclitaxel alone (85 patients), or paclitaxel plus alisertib (84 patients) cohorts.
  *174 women were consented and included in baseline demographics. However, 5 of these did not start study treatment due to ineligibility, participant withdrawal, and/or investigator decision, so only 169 participants were included in Participant Flow and AE/SAE analysis.
Groups:
- ER+/HER2- Paclitaxel Plus Alisertib; Triple Negative Paclitaxel Plus Alisertib: Paclitaxel 60 mg/m2 intravenously (IV) on days 1, 8 and 15 of a 28-day cycle; Alisertib 40 mg BID on days 1-3, 8-10, and 15-17 of a 28-day cycle
  Paclitaxel: either 60 mg/m2 intravenously (IV) on days 1, 8 and 15 of a 28-day cycle (on Paclitaxel plus Alisertib arm) or 90 mg/m2 IV on days 1, 8 and 15 of a 28-day cycle (on Paclitaxel Alone arm)
  Alisertib: 40 mg BID (twice a day) on days 1-3, 8-10, and 15-17 of a 28-day cycle
Period: Overall Study
Arm/Group | ER+/HER2- Paclitaxel Alone | ER+/HER2- Paclitaxel Plus Alisertib | Triple Negative Paclitaxel Alone | Triple Negative Paclitaxel Plus Alisertib
Started | 70 | 66 | 15 | 18
Completed | 36 | 38 | 8 | 10
Not Completed | 34 | 28 | 7 | 8
Not completed — Adverse Event | 13 | 14 | 3 | 2
Not completed — Withdrawal by Subject | 9 | 6 | 3 | 2
Not completed — Physician Decision | 4 | 4 | 0 | 2
Not completed — Other, unrelated complication | 7 | 1 | 1 | 2
Not completed — Death | 1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 174 participants were consented and included in baseline analysis. However, 5 of these did not start study treatment due to ineligibility, participant withdrawal, and/or investigator decision, so only 169 participants were included in Participant Flow and Adverse Event/Serious Adverse Event (AE/SAE) Analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | ER+/HER2- Paclitaxel Alone | ER+/HER2- Paclitaxel Plus Alisertib | Triple Negative Paclitaxel Alone | Triple Negative Paclitaxel Plus Alisertib | Total
Number analyzed (Participants) | 70 | 69 | 16 | 19 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 31 | 4 | 6 | 66
  >=65 years | 45 | 38 | 12 | 13 | 108
Age, Continuous [Median (Full Range); unit: years] | 63.2 [26.9 to 84.2] | 62.5 [33.1 to 83.4] | 65.2 [53.1 to 81.3] | 63.2 [38.8 to 75.0] | 63.2 [26.9 to 84.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 16 | 19 | 174
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 1 | 0 | 3
  Black | 6 | 7 | 6 | 4 | 23
  Caucasian | 55 | 54 | 9 | 13 | 131
  Hispanic | 6 | 6 | 0 | 2 | 14
  Other | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 69 | 16 | 19 | 174
Positive Nodes [Count of Participants; unit: Participants]
  0 | 36 | 33 | 7 | 9 | 85
  1-3 | 20 | 20 | 3 | 4 | 47
  4 or more | 9 | 13 | 5 | 5 | 32
  Missing | 5 | 3 | 1 | 1 | 10
Prior Chemotherapy for Metastatic Disease [Count of Participants; unit: Participants]
  No prior chemotherapy | 48 | 48 | 11 | 13 | 120
  1 prior chemotherapy | 22 | 21 | 5 | 6 | 54
Current Histology [Count of Participants; unit: Participants]
  Ductal | 47 | 45 | 11 | 16 | 119
  Lobular | 10 | 9 | 1 | 0 | 20
  Mixed DL | 2 | 2 | 0 | 0 | 4
  Other | 11 | 13 | 4 | 2 | 30
  Missing | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression - Tumor Response Based on RECIST 1.1 Criteria
Description: Measurement of tumors (sum of longest diameters) every 8 weeks for CT/MRI and photographs, and every 12 weeks for bone scan, if applicable. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions (plus an absolute increase of at least 5 mm), or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death, or discontinuation from study for any other reason, up to 3 years from date of patient registration
Population: All 174 participants who consented were included in this Time to Disease Progression outcome analysis. However, 5 of these participants did not start study treatment, so only 169 participants were included in Safety Analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | ER+/HER2- Paclitaxel Alone | ER+/HER2- Paclitaxel Plus Alisertib | Triple Negative Paclitaxel Alone | Triple Negative Paclitaxel Plus Alisertib
Number analyzed (Participants) | 70 | 69 | 16 | 19
months | 7.1 [3.8 to 10.6] | 10.2 [3.8 to 15.7] | 5.7 [2.9 to 8.2] | 9.6 [6.1 to 22.6]

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause
Time Frame: up to 4 years from date of patient registration
Population: All 174 participants who consented were included in this Overall Survival outcome analysis. However, 5 of these participants did not start study treatment, so only 169 participants were included in Safety Analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ER+/HER2- Paclitaxel Alone | ER+/HER2- Paclitaxel Plus Alisertib | Triple Negative Paclitaxel Alone | Triple Negative Paclitaxel Plus Alisertib
Number analyzed (Participants) | 70 | 69 | 16 | 19
months | 25.1 [16.0 to 30.5] | 26.3 [18.7 to 37.2] | 12.7 [6.8 to 23.5] | 16.0 [9.6 to 34.0]

ADVERSE EVENTS:
Time Frame: until 30 days after last dose of patient's study treatment, for up to 2 years from date of registration (enrollment into study). However, mortality data was collected for up to 4 years from date of registration.
Description: 174 participants consented to study treatment, were randomized and were included in Overall Survival and All-Cause Mortality analysis. However, 5 of these participants did not start study treatment, so only 169 participants were included in AE/SAE Analysis and Participant Flow.
Arm/Group | ER+/HER2- Paclitaxel Alone | ER+/HER2- Paclitaxel Plus Alisertib | Triple Negative Paclitaxel Alone | Triple Negative Paclitaxel Plus Alisertib
All-Cause Mortality (participants affected / at risk) | 43/70 | 39/69 | 14/16 | 13/19
Serious Adverse Events (participants affected / at risk) | 2/70 | 13/66 | 0/15 | 6/18
Other Adverse Events (participants affected / at risk) | 69/70 | 65/66 | 15/15 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ER+/HER2- Paclitaxel Alone (N=70) | ER+/HER2- Paclitaxel Plus Alisertib (N=66) | Triple Negative Paclitaxel Alone (N=15) | Triple Negative Paclitaxel Plus Alisertib (N=18)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
DIARRHEA (Gastrointestinal disorders) | 0 | 3 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 2
INFECTION FUNGAL (Infections and infestations) | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1 | 0 | 0
EMBOLISM PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
INFECTION RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ER+/HER2- Paclitaxel Alone (N=70) | ER+/HER2- Paclitaxel Plus Alisertib (N=66) | Triple Negative Paclitaxel Alone (N=15) | Triple Negative Paclitaxel Plus Alisertib (N=18)
NEUTROPENIA (Blood and lymphatic system disorders) | 13 | 43 | 5 | 14
ANEMIA (Blood and lymphatic system disorders) | 6 | 16 | 5 | 6
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 9 | 2 | 1
HEARTBURN (Cardiac disorders) | 5 | 1 | 0 | 0
EYES TEARING (Eye disorders) | 3 | 1 | 0 | 1
DIARRHEA (Gastrointestinal disorders) | 7 | 39 | 4 | 9
NAUSEA (Gastrointestinal disorders) | 18 | 28 | 6 | 7
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 | 19 | 1 | 4
STOMATITIS (Gastrointestinal disorders) | 7 | 12 | 0 | 2
ANOREXIA (Gastrointestinal disorders) | 6 | 11 | 2 | 1
VOMITING (Gastrointestinal disorders) | 5 | 10 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 11 | 7 | 3 | 6
DYSPEPSIA (Gastrointestinal disorders) | 1 | 5 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4 | 0 | 1
FATIGUE (General disorders) | 27 | 33 | 7 | 9
TASTE ALTERATION (General disorders) | 8 | 5 | 1 | 1
PAIN (General disorders) | 10 | 3 | 1 | 1
EDEMA (General disorders) | 3 | 3 | 0 | 0
EDEMA EXTREMITIES (General disorders) | 5 | 1 | 0 | 1
ALLERGIC REACTION (Immune system disorders) | 3 | 3 | 0 | 1
HYPERSENSITIVITY REACTION (Immune system disorders) | 5 | 0 | 0 | 0
ALT INCREASED (Metabolism and nutrition disorders) | 2 | 6 | 0 | 4 — Elevation of alanine transaminase (ALT) liver enzyme
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 6 | 1 | 3
AST INCREASED (Metabolism and nutrition disorders) | 3 | 4 | 0 | 3 — elevation of aspartate aminotransferase (AST) liver enzyme
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 1
NEUROPATHY (Nervous system disorders) | 7 | 7 | 2 | 0
HEADACHE (Nervous system disorders) | 3 | 6 | 2 | 5
NEUROPATHY PERIPHERAL (Nervous system disorders) | 12 | 4 | 4 | 1
NUMBNESS (Nervous system disorders) | 9 | 3 | 3 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 31 | 31 | 4 | 4
RASH (Skin and subcutaneous tissue disorders) | 5 | 7 | 2 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 7 | 5 | 1 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1

LIMITATIONS AND CAVEATS:
This study has some limitations. First, poor accrual to the TN MBC cohort, likely owing to paclitaxel alone control arm, precludes reliable interpretation of the limited data obtained in this trial. In addition, ER-positive, ERBB2-negative MBC is a heterogeneous disease, and this study does not provide insight into how to identify patients who may benefit from adding alisertib to paclitaxel, as well as those who may not benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT02187991/Prot_SAP_000.pdf